CLINICAL TRIAL: NCT01254955
Title: Antibody Production Following H1N1 Influenza Vaccination in Organ Transplant Patients
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Vanda Friman, MD, PhD, Sahlgrenska University Hospital
Other Study IDs: ALFGBG-141031
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Organ Transplantation
Keywords: 2009 H1N1 influenza vaccine, organ transplant patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- organ transplant patients
  Interventions: Biological: H1N1 vaccine Pandemrix
- healthy controls
  Interventions: Biological: H1N1 vaccine Pandemrix

INTERVENTIONS:
Biological: H1N1 vaccine Pandemrix

SUMMARY:
Organ transplant patients and staff members at the Transplant Institute have received pandemic H1N1 influenza vaccine (Pandemrix) and specific antibody production was measured by haemagglutination inhibition according to the clinical guidelines and policy, respectively. This study retrospectively assessed the immune response after vaccination.

DETAILED DESCRIPTION:
A total of 100 organ transplant patients and 36 healthy controls were included in the study. All individuals were vaccinated between October and November 2009 and received 2 doses of Pandemrix. Serum samples were collected at baseline before vaccination and 1 month after the first and second vaccination. Individual hemagglutination-inhibiting serum antibody titers were measured.Frequency of > 4 -fold increase in antibody titers and seroconversion from non-protective prevaccination titers to protective postvaccination titers were recorded. Adverse events were reported.

ELIGIBILITY:
Inclusion Criteria:

Cohort number 1:Organ transplant patients who were vaccinated and serum sample drawn at baseline.

Cohort number 2: Staff members who were vaccinated and serum sample drawn at baseline.

Exclusion Criteria:

Cohort number 1: Organ transplant patients who were vaccinated and no serum sample drawn at baseline.

Cohort number 2: Staff members who were vaccinated and no serum sample drawn at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tranplant patients at the out-patient clinical ward and staff members at the Transplant Institute, Sahlgrenska University Hospital.
Sampling Method: Probability Sample
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Frequency of responders in organ transplant patients and controls

SECONDARY OUTCOMES:
Frequency of >4-fold titre rise in organ transplant patients and controls

CONTACTS AND LOCATIONS:
Locations (1):
- Transplant Institute, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Result] Felldin M, Studahl M, Svennerholm B, Friman V. The antibody response to pandemic H1N1 2009 influenza vaccine in adult organ transplant patients. Transpl Int. 2012 Feb;25(2):166-71. doi: 10.1111/j.1432-2277.2011.01391.x. Epub 2011 Nov 26. PMID 22117586